CLINICAL TRIAL: NCT00398138
Title: Pilot Trial of a WT-1 Analog Peptide Vaccine in Patients With Thoracic and Myeloid Neoplasms
Brief Title: Vaccine Therapy and GM-CSF in Treating Patients With Acute Myeloid Leukemia, Myelodysplastic Syndromes, Non-Small Cell Lung Cancer, or Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Innovive Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-085; P30CA008748 (NIH); P01CA023766 (NIH); MSKCC-06085
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Leukemia; Lung Cancer; Malignant Mesothelioma; Myelodysplastic Syndromes; Primary Peritoneal Cavity Cancer
Keywords: adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; advanced malignant mesothelioma; recurrent malignant mesothelioma; primary peritoneal cavity cancer
MeSH Terms: conditions — Leukemia; Lung Neoplasms; Mesothelioma, Malignant; Myelodysplastic Syndromes; Congenital Abnormalities; Carcinoma, Non-Small-Cell Lung | interventions — incomplete Freund's adjuvant; sargramostim; Polymerase Chain Reaction; Flow Cytometry; Immunoenzyme Techniques

ARMS (1):
- vaccine (Experimental): Six vaccinations of the WT-1 peptide (1.0 ml of emulsion) will be administered on weeks 0, 4, 6, 8, 10 & 12. Vaccinations will be administered subcutaneously with sites rotated among extremities. Injection sites will be pre-stimulated with Sargramostim (GM-CSF) (70 mcg) injected subcutaneously on days 0 & -2 of each vaccination. Patients may self administer the Sargramostim (GM-CSF) if they have been appropriately instructed on SQ injection administration. Patients will keep a logbook noting the time & placement of the injection. Note: during each vaccination, the Sargramostim (GM-CSF) & the vaccine emulsion will be administered to the same anatomical site. This site will be marked by the patient or treating healthcare professional by a permanent marker pen. For patients who have a clinical, molecular, or immunologic response & have not had disease progression, they may receive up to 6 more vaccinations administered approximately every month.
  Interventions: Biological: WT-1 analog peptide vaccine; Biological: incomplete Freund's adjuvant; Biological: sargramostim; Genetic: polymerase chain reaction; Other: flow cytometry; Other: immunoenzyme technique

INTERVENTIONS:
Biological: WT-1 analog peptide vaccine
Biological: incomplete Freund's adjuvant
Biological: sargramostim
Genetic: polymerase chain reaction
Other: flow cytometry
Other: immunoenzyme technique

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill cancer cells. Biological therapies, such as GM-CSF, may stimulate the immune system in different ways and stop cancer cells from growing. Giving vaccine therapy together with GM-CSF may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects of vaccine therapy and GM-CSF in treating patients with acute myeloid leukemia, myelodysplastic syndromes, non-small cell lung cancer, or mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and immunogenicity of the Wilms tumor-1 analog peptide vaccine in patients with acute myeloid leukemia, myelodysplastic syndromes, non-small cell lung cancer, or mesothelioma.

Secondary

* Determine the antitumor effects of this vaccine in these patients.

OUTLINE: This is a pilot study. Patients are stratified according to disease type (acute myeloid leukemia [AML] or myelodysplastic syndromes [MDS] vs non-small cell lung cancer or mesothelioma).

Patients receive vaccine comprising Wilms-tumor 1 (WT-1) analog peptide emulsified in Montanide ISA-51 subcutaneously (SC) once in weeks 0, 4, 6, 8, 10, and 12 and sargramostim (GM-CSF) SC twice in weeks 0, 4, 6, 8, 10, and 12 (on the day of and 2 days prior to each vaccination). Patients who have an immunologic response and have no disease progression may receive up to 6 more vaccinations approximately 1 month apart.

Blood samples are collected at baseline, week 8, and week 14. Samples are examined by polymerase chain reaction (PCR) to measure levels of WT-1 and by T-cell proliferative response, delayed-type hypersensitivity against WT-1 peptides, or ELISPOT to measure immune response.

Bone marrow samples are collected from patients with AML or MDS at baseline and week 14. Samples are examined by PCR to measure levels of WT-1 and by multiparameter flow cytometry to measure residual disease.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically or histologically confirmed diagnosis of 1 of the following:

  * Acute myeloid leukemia, meeting the following criteria:

    * Documented Wilms tumor-1 (WT-1)-positive disease demonstrated by WT-1 protein on a pretreatment bone marrow biopsy OR detectable disease with real-time quantitative reverse transcriptase-polymerase chain reaction (RQ-PCR)
    * Completed induction chemotherapy, achieved clinical remission, and completed postremission therapy OR achieved clinical remission and have no plans for further postremission chemotherapy (≥ 65 years of age)
  * Myelodysplastic syndromes, meeting the following criteria:

    * Documented WT-1-positive disease demonstrated by WT-1 protein on a pretreatment bone marrow biopsy OR detectable disease by RQ-PCR
    * International Prognostic Scoring System (IPSS) score of ≥ Int-2
    * Not a candidate for cytotoxic chemotherapy
  * Non-small cell lung cancer, meeting the following criteria:

    * Positive tumor staining for WT-1 in > 10% of cells
    * Stage III or IV disease
    * Completed chemotherapy, surgery, and/or radiotherapy
  * Mesothelioma, meeting the following criteria:

    * Positive tumor staining for WT-1 in > 10% of cells
    * Unresectable or relapsed disease
    * Chemo-naive or received 1 prior chemotherapy regimen
    * Malignant pleural mesothelioma or peritoneal mesothelioma
* No leptomeningeal disease
* No CNS involvement

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count > 50,000/mm³ (except for myelodysplastic syndromes where parameter is > 20,000/mm³ and not transfusion dependent)
* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring systemic antibiotics, antiviral, or antifungal treatments
* No serious unstable medical illness

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy or radiotherapy
* No concurrent systemic corticosteroids

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M. Krug, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Maslak PG, Dao T, Krug LM, Chanel S, Korontsvit T, Zakhaleva V, Zhang R, Wolchok JD, Yuan J, Pinilla-Ibarz J, Berman E, Weiss M, Jurcic J, Frattini MG, Scheinberg DA. Vaccination with synthetic analog peptides derived from WT1 oncoprotein induces T-cell responses in patients with complete remission from acute myeloid leukemia. Blood. 2010 Jul 15;116(2):171-9. doi: 10.1182/blood-2009-10-250993. Epub 2010 Apr 16. PMID 20400682
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine: Six vaccinations of the WT-1 peptide (1.0 ml of emulsion) will be administered on weeks 0, 4, 6, 8, 10 & 12. Vaccinations will be administered subcutaneously with sites rotated among extremities. Injection sites will be pre-stimulated with Sargramostim (GM-CSF) (70 mcg) injected subcutaneously on days 0 & -2 of each vaccination. Patients may self administer the Sargramostim (GM-CSF) if they have been appropriately instructed on SQ injection administration. Patients will keep a logbook noting the time & placement of the injection. Note: during each vaccination, the Sargramostim (GM-CSF) & the vaccine emulsion will be administered to the same anatomical site. This site will be marked by the patient or treating healthcare professional by a permanent marker pen. For patients who have a clinical, molecular, or immunologic response & have not had disease progression, they may receive up to 6 more vaccinations administered approximately every month.
  WT-1 analog peptide vaccine
Period: Overall Study
Arm/Group | Vaccine
Started | 12
Completed | 10
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: Toxicities will be tabulated according to the NCI Common Toxicity (version 3.0).
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Vaccine
Number analyzed (Participants) | 10
participants | 10

2. Primary Outcome: Immune Response
Description: Immune reactivity to the peptides will be measured in the same fashion for patients with hematologic or thoracic malignancies. Immune responses will be measured by T cell proliferative response and DTH against WT-1 peptides. In patients with adequate samples, T cell gamma interferon release as measured by ELISPOT will be performed as well.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Vaccine
Number analyzed (Participants) | 10
participants | 10

ADVERSE EVENTS:
Arm/Group | Vaccine
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema: head and neck (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=10)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 10
Hemoglobin (Metabolism and nutrition disorders) | 6
Leukocytes (total WBC) (Infections and infestations) | 4
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Infections and infestations) | 2
Platelets (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes